CLINICAL TRIAL: NCT06533371
Title: Assessment of Pulmonary EmphySema: the Clinical -ULtrasonographic APproach to chronIc Obstructive Pulmonary Disease
Brief Title: Clinical-ultrasonographic Assessment of Pulmonary Emphysema
Acronym: ESCULAPIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Miulli General Hospital (Other); Azienda Ospedaliera di Rilievo Nazionale A.Cardarelli (Other); Università degli Studi di Trento (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 6855; PNRR-MCNT2-2023-12378311 (Other Grant/Funding Number: European Union - Next Generation EU)
Record Dates: First submitted 2024-07-25; First posted 2024-08-01 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Emphysema; Pulmonary Emphysema
Keywords: Pulmonary emphysema; Emphysema; Lung ultrasound; Oscillometry; Quantitative analysis; Chest computed tomography; Early diagnosis
MeSH Terms: conditions — Emphysema; Pulmonary Emphysema; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with pulmonary paraseptal or panlobular emphysema (Experimental): Ultrasonographic findings will be obtained with clinical machines. Additionally, ultrasonographic scans as acquired with research platform will also be gathered.
  LUS findings will be compared to chest computed tomographic findings. Post-processing image analysis of chest CT findings will be performed on images by using automated detection of potential emphysema systems.
  Finally, all COPD patients and subjects who participate in the screening program for lung cancer with CT evidence of paraseptal or panlobular emphysema will undergo respiratory oscillometry.
  Interventions: Diagnostic Test: Relationship between lung ultrasound and computed tomographic scan
- Healthy volunteers and participants without pulmonary emphysema (Experimental): Ultrasonographic findings will be obtained with clinical machines. Additionally, ultrasonographic scans as acquired with research platform will also be gathered.
  LUS findings will be compared to chest computed tomographic findings. Post-processing image analysis of chest CT findings will be performed on images by using automated detection of potential emphysema systems.
  Interventions: Diagnostic Test: Relationship between lung ultrasound and computed tomographic scan

INTERVENTIONS:
Diagnostic Test: Relationship between lung ultrasound and computed tomographic scan — Ultrasonographic findings will be obtained with clinical machines. Additionally, US scans as acquired with the Ula-Op open research platform will also be gathered. For both scanners, 10seconds videos will be recorded and stored in each landmark.
  To correlate LUS artefactual patterns with peripheral parenchymal changes evaluated by HRCT of the chest, all chest CT findings will be analysed by an image processing platform designed to provide visualization and quantification of areas with abnormal CT tissue density indicative of emphysema and air trapping. Post-processing image analysis will be performed on images by using automated detection of potential emphysema systems.

SUMMARY:
The goal of this clinical trial is to identify correlations among data deriving from lung ultrasonographic (LUS) and tomographic evaluations of patients with panlobular or paraseptal emphysema, to improve the comprehension of acoustic information derived from ultrasound evaluation.

The main question it aims to answer is: what are the correlations between thoracic ultrasonographic patterns and peripheral parenchymal changes evaluated by high resolution computed tomography (HRCT) of the chest, in patients affected with variable degree of panlobular or paraseptal emphysema? Researchers will compare LUS patterns observed in: 1) COPD patients with CT evidence of panlobular or paraseptal emphysema, 2) subjects participating in the screening program for lung cancer with CT evidence of panlobular or paraseptal emphysema, and 3) patients with suspected/known lung cancer undergoing with CT evidence of panlobular or paraseptal emphysema, with the ones obtained from healthy volunteers and subjects who participate in the screening program for lung cancer with no evidence of emphysema.

Participants will undergo LUS evaluation with both clinical and research scanners. Patients will be assessed in supine position with the arms extended above the head. The position is the same in which chest CT scans will be performed. LUS assessment will be performed using commercially available linear probes.

Finally, all COPD patients and subjects who participate in the screening program for lung cancer with CT evidence of paraseptal or panlobular emphysema will undergo respiratory oscillometry. Tidal breathing analysis with impulse oscillometry (IOS) has proven to be an informative and meaningful tool used in the early detection and follow up of pulmonary diseases like COPD.

DETAILED DESCRIPTION:
The use of lung ultrasound (LUS) is instrumental in the evaluation of many thoracic diseases and its ability to detect pleural-pulmonary pathologies is widely accepted. However, the use of LUS as an indication of underlying parenchymal lung disease, when the organ is still aerated, is a relatively new application. A-lines and B-lines are two separate and distinct artifacts which may be seen during the examination of the nonconsolidated lungs by ultrasound because of different underlying structures. Even though the practical role of LUS artifacts is accepted for detecting and monitoring many conditions, we do not fully understand their origin. The artifactual information beyond the pleura line in LUS images of the normal and of the not critically deflated lung represents the ultimate outcome of complex interactions of a specific acoustic wave with a specific three-dimensional structure of the biological tissue.

Chronic obstructive pulmonary disease (COPD) is a complex condition with a wide spectrum of clinical presentations and pathological features unified under the spirometric definition of airflow obstruction. The mechanisms responsible for airflow obstruction in COPD (airway narrowing and parenchymal destruction) cannot be distinguished by standard spirometry.

Chest computed tomography (CT) allows to depict and measure in vivo the lung pathologic changes of COPD by quantifying parenchymal destruction, the direct sign of emphysema. Although quantitative and qualitative studies have shown that CT can allow distinguishing subtypes of emphysema, a widespread routine use of CT for the assessment of COPD in clinical practice cannot be currently foreseen due to radiation exposure and limited instrumental availability.

LUS can detect pleural-pulmonary pathologies. However, the use of LUS as an indication of underlying parenchymal lung disease, when the organ is still aerated, as in emphysema, is a new application.

This study is aimed at researching correlations among a pool of data deriving from ultrasonographic and tomographic evaluations of patients with panlobular or paraseptal emphysema, to improve the comprehension of acoustic information derived from ultrasound evaluation.

The study will not modify the diagnostic / therapeutic process of the enrolled patients, who will all have in common the CT evidence of panlobular or paraseptal emphysema.

Researchers will observe three defined population of patients at a single point (at the time of enrolment). All subjects will have CT evidence of panlobular or paraseptal emphysema. Patients will be recruited through three paths: 1) patients suffered from COPD, in follow-up at Pulmonary Medicine Units in Rome and Naples, with HRCT evidence of paraseptal or panlobular emphysema; 2) subjects who participate in the screening program for lung cancer in Rome, Naples and Acquaviva delle Fonti, and 3) patients with suspected/known lung cancer managed in all medical Units involved in this project.

All enrolled subjects will undergo LUS evaluation with both clinical and research scanners. Patients will be assessed in supine position with the arms extended above the head. The position is the same in which chest CT scans will be performed. LUS assessment will be performed using commercially available linear probes.

Finally, all COPD patients and subjects who participate in the screening program for lung cancer with CT evidence of paraseptal or panlobular emphysema will undergo oscillometry. Tidal breathing analysis with impulse oscillometry (IOS) has proven to be an informative and meaningful tool used in the early detection and follow up of pulmonary diseases like COPD. IOS is almost independent of patient cooperation and can test a larger patient range than spirometry alone including geriatric patients.

ELIGIBILITY:
Inclusion Criteria:

* outpatients in follow-up for chronic obstructive pulmonary disease, in stable conditions, with computed tomographic evidence of panlobular or paraseptal emphysema.
* Inpatients, admitted to the hospital due to acute exacerbation of chronic obstructive pulmonary disease, with computed tomographic evidence of panlobular or paraseptal emphysema.
* Subjects who participate in the screening program for lung cancer with computed tomographic evidence of panlobular or paraseptal emphysema.
* Outpatients / Inpatients with suspected/known lung cancer and computed tomographic evidence of panlobular or paraseptal emphysema.
* Patients able to give written informed consent.

Exclusion Criteria:

* pregnancy.
* Pediatric population.
* Patients unable to express written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1628 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with ultrasonographic pattern of emphysema. | through study completion, an average of 2 year
  To characterize ultrasonographic signs of paraseptal or panlobular emphysema, the measurement of the ultrasound backscattering-index, as a function of the transmitted frequency, will be perform.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Inchingolo, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (4):
- Italy (4):
  - Ente Ecclesiastico, Ospedale Generale Regionale "F. Miulli", Acquaviva delle Fonti
  - A.O.R.N. "A. Cardarelli", Napoli
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
  - University of Trento, Trento

IPD SHARING:
Plan to Share IPD: No
Researchers intend to communicate the trial results to participants, healthcare professionals, and other relevant groups through scientific publications and national and international conference proceedings. No individual participant data will be available.
  Any document produced, including scientific publications relating to the research project will contain an explicit indication that the project is financed under the PNRR statement stating "funded by the European Union - Next Generation EU - PNRR M6C2 - Investment 2.1 Enhancement and strengthening of biomedical research in the NHS", the emblem of the Union European Union and the project code. The products will be made public through systems that allow immediate use by the public (for example open-access).

REFERENCES:
- [Background] Mento F, Perini M, Malacarne C, Demi L. Ultrasound multifrequency strategy to estimate the lung surface roughness, in silico and in vitro results. Ultrasonics. 2023 Dec;135:107143. doi: 10.1016/j.ultras.2023.107143. Epub 2023 Aug 24. PMID 37647701
- [Background] Wolfram F, Miller D, Demi L, Verma P, Moran CM, Walther M, Mathis G, Prosch H, Kollmann C, Jenderka KV. Best Practice Recommendations for the Safe use of Lung Ultrasound. Ultraschall Med. 2023 Oct;44(5):516-519. doi: 10.1055/a-1978-5575. Epub 2022 Nov 14. PMID 36377189
- [Background] Demi L, Wolfram F, Klersy C, De Silvestri A, Ferretti VV, Muller M, Miller D, Feletti F, Welnicki M, Buda N, Skoczylas A, Pomiecko A, Damjanovic D, Olszewski R, Kirkpatrick AW, Breitkreutz R, Mathis G, Soldati G, Smargiassi A, Inchingolo R, Perrone T. New International Guidelines and Consensus on the Use of Lung Ultrasound. J Ultrasound Med. 2023 Feb;42(2):309-344. doi: 10.1002/jum.16088. Epub 2022 Aug 22. PMID 35993596
- [Background] Mento F, Khan U, Faita F, Smargiassi A, Inchingolo R, Perrone T, Demi L. State of the Art in Lung Ultrasound, Shifting from Qualitative to Quantitative Analyses. Ultrasound Med Biol. 2022 Dec;48(12):2398-2416. doi: 10.1016/j.ultrasmedbio.2022.07.007. Epub 2022 Sep 23. PMID 36155147
- [Background] Mento F, Demi L. Dependence of lung ultrasound vertical artifacts on frequency, bandwidth, focus and angle of incidence: An in vitro study. J Acoust Soc Am. 2021 Dec;150(6):4075. doi: 10.1121/10.0007482. PMID 34972265
- [Background] Guidi F, Demi L, Tortoli P. Experimental and simulation study of harmonic components generated by plane and focused waves. Ultrasonics. 2021 Sep;116:106504. doi: 10.1016/j.ultras.2021.106504. Epub 2021 Jun 22. PMID 34216989
- [Background] Peschiera E, Mento F, Demi L. Numerical study on lung ultrasound B-line formation as a function of imaging frequency and alveolar geometries. J Acoust Soc Am. 2021 Apr;149(4):2304. doi: 10.1121/10.0003930. PMID 33940883
- [Background] Mento F, Demi L. On the influence of imaging parameters on lung ultrasound B-line artifacts, in vitro study. J Acoust Soc Am. 2020 Aug;148(2):975. doi: 10.1121/10.0001797. PMID 32873037
- [Background] Soldati G, Demi M, Smargiassi A, Inchingolo R, Demi L. The role of ultrasound lung artifacts in the diagnosis of respiratory diseases. Expert Rev Respir Med. 2019 Feb;13(2):163-172. doi: 10.1080/17476348.2019.1565997. Epub 2019 Jan 10. PMID 30616416
- [Background] Occhipinti M, Paoletti M, Bartholmai BJ, Rajagopalan S, Karwoski RA, Nardi C, Inchingolo R, Larici AR, Camiciottoli G, Lavorini F, Colagrande S, Brusasco V, Pistolesi M. Spirometric assessment of emphysema presence and severity as measured by quantitative CT and CT-based radiomics in COPD. Respir Res. 2019 May 23;20(1):101. doi: 10.1186/s12931-019-1049-3. PMID 31122243
- [Background] Occhipinti M, Paoletti M, Bigazzi F, Camiciottoli G, Inchingolo R, Larici AR, Pistolesi M. Emphysematous and Nonemphysematous Gas Trapping in Chronic Obstructive Pulmonary Disease: Quantitative CT Findings and Pulmonary Function. Radiology. 2018 May;287(2):683-692. doi: 10.1148/radiol.2017171519. Epub 2018 Jan 23. PMID 29361243
- [Background] Veneroni C, Gobbi A, Pompilio PP, Dellaca R, Fasola S, La Grutta S, Leyva A, Porszasz J, Stornelli SR, Fuso L, Valach C, Breyer-Kohansal R, Breyer MK, Hartl S, Contu C, Inchingolo R, Hodgdon K, Kaminsky DA. Reference Equations for Within-Breath Respiratory Oscillometry in White Adults. Respiration. 2024;103(9):521-534. doi: 10.1159/000539532. Epub 2024 Jun 7. PMID 38843786